CLINICAL TRIAL: NCT03462732
Title: Nasotracheal Tube Stenting by Nelaton Catheter in Pediatric Dental Surgery , Prospective Randomized Clinical Trial
Brief Title: Nasotracheal Tube Stenting by Nelaton Catheter in Pediatric Dental Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amin Mohammed Alansary Amin Ahmed Helwa, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FAMSU R 6 / 2018
Record Dates: First submitted 2018-02-24; First posted 2018-03-13 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Anesthesia Intubation Complication
MeSH Terms: interventions — Stents

STUDY DESIGN:
Intervention Model Description: assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): Endotracheal tube plus Nelaton catheter
  Interventions: Device: Endotracheal tube; Device: Nelaton catheter
- Group II (Active Comparator): Endotracheal tube
  Interventions: Device: Endotracheal tube

INTERVENTIONS:
Device: Endotracheal tube — Nasotracheal intubation will be done with endotracheal tube
Device: Nelaton catheter — plus nelaton catheter
  Other Names: Stent
  Arms: Group I

SUMMARY:
The value of this study is to compare between stented endotracheal tube with nelaton catheter and non stented tube as regard nasotracheal related complications as epistaxis and nasal cavity injury.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients scheduled for dental surgery under general anesthesia age 3-9 years
* physical status American society of Anesthesiologist(ASA) I orII

Exclusion Criteria:

* History of recurrent epistaxis
* Coagulopathy
* Previous nasal surgery
* History of nasal trauma
* Severe renal , hepatic or cardiovascular disease
* History of drug allergy to the drugs used in the study

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
incidence and severity of Epistaxis | immediately after nasotracheal intubation
  An independent anesthesiologist who did not observe the tube insertion will assess the incidence and severity of epistaxis using a laryngoscope immediately after tube passage through the nasal cavity , four grades to evaluate epistaxis 1- no epistaxis 2- mild epistaxis ,blood apparent on the surface of the tube 3-moderate epistaxis pooling of blood on the posterior pharyngeal wall 4- severe epistaxis , large amount of blood in the pharynx impeding nasotracheal intubation and necessitating urgent orotracheal intubation.

SECONDARY OUTCOMES:
Histopathology of the endotracheal tube contents after extubation | immediately after extubation
  after extubation the tube contents will be collected in a 5 ml syringe by using sterile swab then tissues will be separated and will be sent for histopathology , the remnant contents will be sent for microscopy , grading the contents as follow 1- secretions only 2- secretions plus blood 3- secretions , blood plus tissues .

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided